CLINICAL TRIAL: NCT02951819
Title: Daratumumab Plus Cyclophosphamide, Bortezomib and Dexamethasone (Dara-CyBorD) in Previously Untreated and Relapsed Subjects With Multiple Myeloma
Brief Title: A Study to Evaluate Dara-CyBorD in Previously Untreated and Relapsed Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108235; 54767414MMY2012 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Cyclophosphamide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Dara-CyBorD (Experimental): Subjects will receive Daratumumab along with Cyclophosphamide, Bortezomib and Dexamethasone (Dara-CyBorD) as induction on a 28-day cycle length and Daratumab and Dexamethasone on Day 1 of each cycle for 12 cycles as maintenance therapy.
  Interventions: Drug: Daratumumab; Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — For induction therapy cycle 1 day 1 and day 2 doses of daratumumab will be 8 milligram/kilogram (mg/kg). Starting cycle 1 week 2 until the completion of week 8 of daratumumab patients will receive 16 mg/kg Intravenously (IV) weekly.
  Starting week 9 until the completion of week 24 therapy daratumumab will be administered every other week at 16 mg/kg IV.
  Starting week 25 and beyond for induction therapy daratumumab will be given once every 4 weeks.
Drug: Cyclophosphamide — Subjects will receive 4 to 8 cycles of oral cyclophosphamide 300 milligram per meter square (mg/m^2 ) on Days 1, 8, 15, and 22 for every 28 days.
Drug: Bortezomib — Subjects will receive 4 to 8 cycles of Bortezomib 1.5 mg/m2 subcutaneous (SC) on Days 1, 8, and 15 for every 28 days.
Drug: Dexamethasone — Subjects will be given corticosteroids (Dexamethasone) as pre-infusion therapy prior to daratumumab and for the first 8 cycles will also receive post-infusion corticosteroids (Dexamethasone).

SUMMARY:
The purpose of this study is to evaluate complete response plus (+) very good partial response (CR+VGPR) rate following 4 cycles of induction therapy of daratumumab in combination with cyclophosphamide, bortezomib, and dexamethasone (Dara-CyBorD), in previously untreated subjects, and in relapsed subjects with multiple myeloma, as defined by the International Myeloma Working Group (IMWG) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented multiple myeloma (MM) as defined by the International Myeloma Working Group (IMWG) 2015 criteria: Clonal bone marrow plasma cells greater than or equal to (>=) 10 percent (%) or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following CRAB (calcium level, renal dysfunction, anemia, and destructive bone lesions) features and myeloma defining events as in the protocol
* Subjects with previously untreated myeloma or relapsed myeloma with one prior line of therapy including an induction regimen which may be followed by autologous stem cell transplantation and single agent maintenance therapy. For previously untreated subjects an emergency course of steroids (defined as no greater than 40 milligram (mg) of dexamethasone, or equivalent per day for a maximum of 4 days) is permitted. In addition, radiation therapy is permitted prior to study entry, during screening, and during Cycles 1-2 of study treatment as needed for lytic bone disease
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* A woman of childbearing potential must have 2 negative serum (beta (β) human chorionic gonadotropin) or urine pregnancy tests during screening, the first one within 28 days prior to the first dose of study drug and the second within 24 hours prior to the first dose of study drug
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control example, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Refractory to any proteasome inhibitor (PI) or the combination of PI and immunomodulatory drug (IMiD) agents (such as lenalidomide), defined as failure to respond or progression within 60 days of the end of PI therapy
* Exhibiting clinical signs of or has a known history of meningeal or central nervous system involvement by multiple myeloma
* Has known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) less than (<) 50 percent (%) of predicted normal
* Has known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification
* Is known to be seropositive for human immunodeficiency virus, known to have hepatitis B surface antigen positivity, or known to have a history of hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2020-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (26):
- United States (26):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Sedona, Arizona
  - Tucson, Arizona
  - Fayetteville, Arkansas
  - Greenbrae, California
  - Denver, Colorado
  - Niles, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Bethesda, Maryland
  - Columbia, Maryland
  - Grand Rapids, Michigan
  - Omaha, Nebraska
  - Camden, New Jersey
  - Albany, New York
  - East Setauket, New York
  - Fresh Meadows, New York
  - Cincinnati, Ohio
  - Eugene, Oregon
  - Greenville, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Seattle, Washington

REFERENCES:
- [Derived] Yimer H, Melear J, Faber E, Bensinger WI, Burke JM, Narang M, Stevens D, Gray KS, Lutska Y, Bobba P, Qi K, Hoehn D, Qi M, Lin TS, Rifkin RM. Daratumumab, cyclophosphamide, bortezomib, and dexamethasone for multiple myeloma: final results of the LYRA study. Leuk Lymphoma. 2022 Oct;63(10):2383-2392. doi: 10.1080/10428194.2022.2076847. Epub 2022 Jun 22. PMID 35730586

RESULTS

PARTICIPANT FLOW:
Groups:
- Newly Diagnosed Multiple Myeloma (NDMM): Induction therapy:Participants received daratumumab, cyclophosphamide, bortezomib, and dexamethasone (Dara-CyBorD) as: daratumumab 8 mg/kg IV on Cycle 1(Day 1,2) and 16 mg/kg IV on Cycle 1(Days 8,15,22), Cycle 2 (Days 1,8,15,22), Cycles 3-6 (Days 1,15), Cycles 7-8(Day 1); Cyclophosphamide 300 mg/m^2 orally on Days 1,8,15,22 of each cycle (28 days); Bortezomib 1.5 mg/m^2 SC on Days 1,8,15 of each cycle; Dexamethasone 20 mg IV on Cycle 1(Day1,2,8,15,22) and orally on Cycle 1(Day 9,16,23), 40 mg IV or oral on Cycle 2 (Days 1,8,15,22), Cycle 3-8 ([if with CyBorD] Days 1,8,15,22). Consolidation therapy (CT): Participants who were considered eligible for transplant underwent autologous stem cell transplantation [ASCT] at investigator discretion. Maintenance therapy: Daratumumab 16 mg/kg IV on Day 1 for 12 cycles or until PD, whichever occurred first; Dexamethasone 12 mg IV or oral on Day 1 of each cycle(for ASCT participants, maintenance therapy was to begin approximately 90 days after ASCT).
- Relapsed Multiple Myeloma (RMM): Participants with RMM (defined as having achieved at least a PR with first-line therapy before progression) received treatment as-Induction therapy:Participants received Dara-CyBorD as: daratumumab 8 mg/kg IV on Cycle 1(Day 1,2) and 16 mg/kg IV on Cycle 1(Days 8,15,22),Cycle 2 (Days 1,8,15,22),Cycles 3-6(Days 1,15),Cycles 7-8(Day 1); Cyclophosphamide 300 mg/m^2 orally on Days 1,8,15,22 of each cycle (28 days); Bortezomib 1.5 mg/m^2 SC on Days 1,8,15 of each cycle; Dexamethasone 20 mg IV on Cycle 1(Day1,2,8,15,22) and orally on Cycle 1(Day 9,16,23), 40 mg IV or oral on Cycle 2(Days 1,8,15,22),Cycle 3-8 ([if with CyBorD] Days 1,8,15,22). CT: Participants who were considered eligible for transplant underwent ASCT at investigator discretion. Maintenance therapy: Daratumumab 16 mg/kg IV on Day 1 for 12 cycles or until PD, whichever occurred first; Dexamethasone 12 mg IV or oral on Day 1 of each cycle(for ASCT participants, maintenance therapy was to begin approximately 90 days after ASCT).
Period: Overall Study
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Started | 87 | 14
Treated | 86 | 14
Completed | 59 | 7
Not Completed | 28 | 7
Not completed — Death | 9 | 7
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Progressive Disease | 1 | 0
Not completed — Other | 9 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included enrolled participants who received at least 1 dose (partial or complete) of study treatment (Dara-CyBorD).
Groups:
- Total: Total of all reporting groups
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM) | Total
Number analyzed (Participants) | 86 | 14 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9) | 66.4 (8.97) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 4 | 36
  Male | 54 | 10 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 79 | 12 | 91
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 0 | 11
  White | 67 | 14 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 0 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 86 | 14 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Complete Response (CR) or Very Good Partial Response (VGPR)
Description: Percentage of participants who achieved CR or VGPR (as per International Myeloma Working Group [IMWG] criteria) was reported. CR: negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and less than (<) 5 percent (%) plasma cells (PC) in bone marrow. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or greater than or equal to (>=) 90% reduction in serum M-protein plus urine M-protein level < 100 milligram per 24 hours (mg/24hours).
Time Frame: After 4 cycles of Induction (Approximately 4 months)
Population: Response-evaluable set includes all enrolled participants who had measurable disease, received at least 1 dose of study treatment, and had at least 1 efficacy evaluation assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Newly Diagnosed Multiple Myeloma (NDMM): Induction therapy:Participants received daratumumab, cyclophosphamide, bortezomib, and dexamethasone (Dara-CyBorD) as: daratumumab 8 mg/kg IV on Cycle 1(Day 1,2) and 16 mg/kg IV on Cycle 1(Days 8,15,22), Cycle 2 (Days 1,8,15,22), Cycles 3-6 (Days 1,15), Cycles 7-8(Day 1); Cyclophosphamide 300 mg/m^2 orally on Days 1,8,15,22 of each cycle (28 days); Bortezomib 1.5 mg/m^2 SC on Days 1,8,15 of each cycle; Dexamethasone 20 mg IV on Cycle 1(Day1,2,8,15,22) and orally on Cycle 1(Day 9,16,23), 40 mg IV or oral on Cycle 2 (Days 1,8,15,22), Cycle 3-8 ([if with CyBorD] Days 1,8,15,22). Consolidation therapy (CT):Participants who were considered eligible for transplant underwent autologous stem cell transplantation [ASCT] at investigator discretion. Maintenance therapy:Daratumumab 16 mg/kg IV on Day 1 for 12 cycles or until PD, whichever occurred first; Dexamethasone 12 mg IV or oral on Day 1 of each cycle(for ASCT participants, maintenance therapy was to begin approximately 90 days after ASCT).
- Relapsed Multiple Myeloma (RMM): Participants with RMM (defined as having achieved at least a PR with first-line therapy before progression) received treatment as-Induction therapy:Participants received Dara-CyBorD as: daratumumab 8 mg/kg IV on Cycle 1(Day 1,2) and 16 mg/kg IV on Cycle 1(Days 8,15,22),Cycle 2 (Days 1,8,15,22),Cycles 3-6(Days 1,15),Cycles 7-8(Day 1); Cyclophosphamide 300 mg/m^2 orally on Days 1,8,15,22 of each cycle (28 days); Bortezomib 1.5 mg/m^2 SC on Days 1,8,15 of each cycle; Dexamethasone 20 mg IV on Cycle 1(Day1,2,8,15,22) and orally on Cycle 1(Day 9,16,23), 40 mg IV or oral on Cycle 2(Days 1,8,15,22),Cycle 3-8 ([if with CyBorD] Days 1,8,15,22). CT: Participants who were considered eligible for transplant underwent ASCT at investigator discretion. Maintenance therapy:Daratumumab 16 mg/kg IV on Day 1 for 12 cycles or until PD, whichever occurred first; Dexamethasone 12 mg IV or oral on Day 1 of each cycle(for ASCT participants, maintenance therapy was to begin approximately 90 days after ASCT).
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 86 | 14
Percentage of Participants | 44.2 [33.5 to 55.3] | 57.1 [28.9 to 82.3]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR: percentage of participants achieved PR or better (PR,VGPR,CR,sCR) per IMWG. CR:negative immunofixation on serum, urine, disappearance of soft tissue plasmacytomas,<5% PCs in bone marrow(BM). sCR:CR plus normal FLC ratio,absence of clonal cells in BM by immunohistochemistry, immunofluorescence. VGPR:Serum, urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein plus urine M-protein level <100 mg/24hours. PR:>=50% reduction of serum M-protein and reduction in 24hours urinary M-protein by >=90% or to <200mg/24hours. If serum, urine M-protein unmeasurable, a>=50% decrease in difference involved and uninvolved FLC levels required in place of M-protein criteria. If serum, urine M-protein not measurable, serum free light assay is not measurable,>=50% reduction in PCs required in place of M-protein,provided baseline bone marrow PCs% >=30%, if present at baseline, a >=50% reduction in size of soft tissue plasmacytomas is also required.
Time Frame: After 4 Cycles of Induction (4 months), at End of Induction (4 to 8 months) and at the End of Maintenance (12 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 86 | 14
Percentage of participants
  After 4 Cycles of Induction | 79.1 [69.0 to 87.1] | 71.4 [41.9 to 91.6]
  At the End of Induction | 87.2 [78.3 to 93.4] | 78.6 [49.2 to 95.3]
  At the End of Maintenance | 89.5 [81.1 to 95.1] | 85.7 [57.2 to 98.2]

3. Secondary Outcome: Time to Very Good Partial Response (VGPR) or Better
Description: Time to VGPR or Better response was defined as duration from the date of first dose (start of induction) to the date of initial documentation of the response (VGPR or better) which was confirmed by a repeated measurement as required by the IMWG criteria. VGPR is defined by IMWG criteria as serum and urine M-protein detectable by immunofixation but not on electrophoresis or greater than or equal to (>=) 90 % reduction in serum M-protein plus urine M-protein level < 100 milligram/24 hours (mg/24 hours).
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 86 | 14
Months | 3.8 [2.8 to 4.9] | 1.8 [1.0 to 4.7]

4. Secondary Outcome: Time to Partial Response (PR) or Better
Description: Time to PR or Better response was defined as duration from the date of first dose (start of induction) to the date of initial documentation of the response (PR or better) which was confirmed by a repeated measurement as required by the IMWG criteria. PR is defined as per IMWG criteria as >= 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >= 90% or to < 200 mg/24hours. If the serum and urine M-protein are unmeasurable, a>= 50% decrease in the difference between involved and uninvolved Free light chain (FLC) levels is required in the place of the M-protein criteria. If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cells percentage was >=30%. In addition to the above listed criteria, if present at baseline, a >= 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 86 | 14
Months | 1.0 [1.0 to 1.0] | 1.0 [0.9 to 7.4]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined for participants with a confirmed response (PR or better) as the duration from the date of initial documentation of a response (PR or better) according to the IMWG criteria to the date of first documented evidence of progressive disease according to the IMWG criteria or death due to progressive disease. PR:>=50% reduction of serum M-protein and reduction in 24hours urinary M-protein by >=90% or to <200 mg/24hours. If serum and urine M-protein are unmeasurable, a >=50% decrease in difference involved and uninvolved FLC levels required in place of M-protein criteria. If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in PCs is required in place of M-protein, provided baseline bone marrow PCs % was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Up to 36 months
Population: Population included responders (PR or better) in response-evaluable set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 77 | 12
Months | NA [NA to NA] — NA indicates that the median, lower and upper limit of confidence interval (CI) was not estimable due to insufficient number of events to determine this value. | 20.7 [5.9 to NA] — NA indicates that the upper limit of CI was not estimable due to insufficient number of events to determine this value.

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS: duration from date of first dose (start of induction) to date of first documented evidence of progressive disease (PD) based on computerized algorithm per IMWG criteria or death due to any cause, whichever occurred first. PD: 25% increase from lowest response value in one of following: Serum and urine M-component (absolute increase >=0.5 g/dL and >=200 mg/24 hours respectively);Only participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase>10 mg/dL);Only participants without measurable serum and urine M-protein levels, without measurable disease by FLC levels, bone marrow PC% (absolute % >=10%); Bone marrow PC%: absolute% >10%; Definite development of new bone lesions/soft tissue plasmacytomas/definite increase in size of existing bone lesions/soft tissue plasmacytomas, Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: Up to 36 months
Population: Full analysis set is defined as enrolled participants who provided informed consent and met eligibility criteria.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 87 | 14
Months | NA [NA to NA] — NA indicates that the median, lower and upper limit of CI was not estimable due to insufficient number of events to determine this value. | 21.7 [6.8 to NA] — NA indicates that the upper limit of CI was not estimable due to insufficient number of events to determine this value.

7. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP was defined as the time between the date of first dose (start of induction) and the date of first documented evidence of confirmed PD, as defined in the IMWG response criteria. PD per IMWG criteria: Increase of 25% from lowest response value in one of following: Serum and urine M-component (absolute increase >=0.5 g/deciliter (dL) and >=200 mg/24 hours respectively); Only participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase>10 mg/dL); Only participants without measurable serum and urine M-protein levels, without measurable disease by FLC levels, bone marrow PC% (absolute % >=10%); Bone marrow PC%: absolute% >10%; Definite development of new bone lesions/soft tissue plasmacytomas/definite increase in size of existing bone lesions/soft tissue plasmacytomas and Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the PC proliferative disorder.
Time Frame: Approximately 15 months
Population: Full Analysis Set defined as enrolled subjects who provided informed consent and met eligibility criteria.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 87 | 14
Months | NA [NA to NA] — NA indicates that the median, lower and upper limit of CI was not estimable due to insufficient number of events to determine this value. | 13.31 [6.80 to 13.31]

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was measured from the date of first dose (start of induction) to the date of death due to any cause.
Time Frame: Up to 36 months
Population: Full analysis set is defined as enrolled participants who provided informed consent and met eligibility criteria.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 87 | 14
Months | NA [NA to NA] — NA indicates that median, lower and upper limit of CI was not estimable due to insufficient number of events to determine this value. | NA [11.30 to NA] — NA indicates that median and upper limit of CI was not estimable due to insufficient number of events to determine this value.

9. Secondary Outcome: Percentage of Participants With Treatment Emergent-Adverse Event
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between administration of study drug and approximately up to 36 months that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Up to 36 months
Population: Safety Analysis Set defined as enrolled participants who received at least 1 dose (partial or complete) of study treatment (Dara-CyBorD).
Measure: Number; unit: Percentage of participants
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
Number analyzed (Participants) | 86 | 14
Percentage of participants | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Up to 36 months
Description: Safety analysis set is defined as enrolled participants who received at least 1 dose (partial or complete) of study treatment (Dara-CyBorD).
Arm/Group | Newly Diagnosed Multiple Myeloma (NDMM) | Relapsed Multiple Myeloma (RMM)
All-Cause Mortality (participants affected / at risk) | 9/86 | 7/14
Serious Adverse Events (participants affected / at risk) | 28/86 | 5/14
Other Adverse Events (participants affected / at risk) | 86/86 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Newly Diagnosed Multiple Myeloma (NDMM) (N=86) | Relapsed Multiple Myeloma (RMM) (N=14)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 4 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial Sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Herpes Zoster Disseminated (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia Parainfluenzae Viral (Infections and infestations) | 1 | 0
Pneumonia Streptococcal (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Newly Diagnosed Multiple Myeloma (NDMM) (N=86) | Relapsed Multiple Myeloma (RMM) (N=14)
Anaemia (Blood and lymphatic system disorders) | 12 | 1
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 1
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 8 | 2
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2
Atrial Fibrillation (Cardiac disorders) | 4 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 3 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Deafness Bilateral (Ear and labyrinth disorders) | 1 | 0
Ear Congestion (Ear and labyrinth disorders) | 2 | 0
Ear Discomfort (Ear and labyrinth disorders) | 2 | 0
Ear Pain (Ear and labyrinth disorders) | 2 | 0
Eustachian Tube Obstruction (Ear and labyrinth disorders) | 0 | 1
Excessive Cerumen Production (Ear and labyrinth disorders) | 2 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 4 | 0
Cataract Subcapsular (Eye disorders) | 1 | 0
Chalazion (Eye disorders) | 2 | 0
Diplopia (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 4 | 0
Eye Discharge (Eye disorders) | 0 | 1
Eye Irritation (Eye disorders) | 2 | 0
Eye Pruritus (Eye disorders) | 1 | 0
Eye Swelling (Eye disorders) | 1 | 0
Lacrimation Increased (Eye disorders) | 4 | 2
Ocular Hyperaemia (Eye disorders) | 1 | 0
Periorbital Oedema (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 2 | 0
Retinal Haemorrhage (Eye disorders) | 1 | 0
Swelling of Eyelid (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 4 | 2
Visual Impairment (Eye disorders) | 0 | 1
Vitreous Floaters (Eye disorders) | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 8 | 4
Abdominal Pain Lower (Gastrointestinal disorders) | 3 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 0
Anal Incontinence (Gastrointestinal disorders) | 1 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 27 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0
Dental Discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 38 | 6
Diverticulum (Gastrointestinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 10 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 2
Gingival Disorder (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hyperaesthesia Teeth (Gastrointestinal disorders) | 1 | 0
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 43 | 3
Oesophageal Pain (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 1
Oral Pain (Gastrointestinal disorders) | 2 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1
Swollen Tongue (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 6 | 0
Vomiting (Gastrointestinal disorders) | 25 | 5
Vomiting Projectile (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 3 | 1
Axillary Pain (General disorders) | 2 | 0
Catheter Site Bruise (General disorders) | 1 | 0
Catheter Site Erythema (General disorders) | 1 | 0
Catheter Site Haemorrhage (General disorders) | 1 | 0
Catheter Site Pain (General disorders) | 2 | 0
Catheter Site Pruritus (General disorders) | 1 | 0
Chest Discomfort (General disorders) | 6 | 2
Chest Pain (General disorders) | 2 | 0
Chills (General disorders) | 17 | 1
Face Oedema (General disorders) | 2 | 0
Fatigue (General disorders) | 58 | 7
Feeling Cold (General disorders) | 2 | 0
Feeling Hot (General disorders) | 0 | 1
Feeling Jittery (General disorders) | 0 | 1
Gait Disturbance (General disorders) | 1 | 1
Influenza Like Illness (General disorders) | 2 | 1
Infusion Site Extravasation (General disorders) | 1 | 1
Injection Site Erythema (General disorders) | 3 | 1
Injection Site Pain (General disorders) | 1 | 0
Injection Site Rash (General disorders) | 1 | 1
Injection Site Reaction (General disorders) | 4 | 0
Localised Oedema (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Medical Device Discomfort (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 4 | 0
Oedema (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 21 | 1
Pain (General disorders) | 6 | 2
Peripheral Swelling (General disorders) | 1 | 2
Pyrexia (General disorders) | 17 | 1
Tenderness (General disorders) | 0 | 1
Thirst (General disorders) | 1 | 0
Xerosis (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 2 | 1
Hypogammaglobulinaemia (Immune system disorders) | 2 | 1
Seasonal Allergy (Immune system disorders) | 6 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0
Arthritis Infective (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 7 | 1
Bronchitis Viral (Infections and infestations) | 2 | 0
Candida Infection (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 6 | 0
Cytomegalovirus Chorioretinitis (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Ear Infection (Infections and infestations) | 1 | 0
Eye Infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 2 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Gingival Abscess (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Herpes Zoster Disseminated (Infections and infestations) | 2 | 0
Hordeolum (Infections and infestations) | 11 | 0
Infected Bite (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 6 | 0
Localised Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 11 | 5
Oral Candidiasis (Infections and infestations) | 1 | 0
Oral Herpes (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 3
Pseudomonal Bacteraemia (Infections and infestations) | 0 | 1
Rash Pustular (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 7 | 4
Skin Infection (Infections and infestations) | 2 | 0
Tinea Infection (Infections and infestations) | 1 | 0
Tooth Abscess (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 30 | 7
Urinary Tract Infection (Infections and infestations) | 7 | 0
Viral Infection (Infections and infestations) | 3 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Wound Infection (Infections and infestations) | 1 | 0
Abdominal Wall Wound (Injury, poisoning and procedural complications) | 1 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1
Bone Contusion (Injury, poisoning and procedural complications) | 1 | 0
Bone Fragmentation (Injury, poisoning and procedural complications) | 1 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 1
Eye Contusion (Injury, poisoning and procedural complications) | 0 | 1
Eyelid Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 10 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 3 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 3 | 0
Radiation Skin Injury (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 5 | 0
Aspartate Aminotransferase Increased (Investigations) | 6 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 2 | 0
Blood Creatinine Increased (Investigations) | 5 | 1
Blood Pressure Increased (Investigations) | 1 | 1
Breath Sounds Abnormal (Investigations) | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 0
Oxygen Saturation Decreased (Investigations) | 2 | 1
Prostatic Specific Antigen Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 7 | 0
Weight Increased (Investigations) | 8 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 18 | 2
Dehydration (Metabolism and nutrition disorders) | 15 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 2 | 0
Fluid Retention (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 27 | 6
Bone Lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 10 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Extremity Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 5 | 1
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8 | 1
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 9 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 12 | 3
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Myalgia Intercostal (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 15 | 4
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 3 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urethral Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anosmia (Nervous system disorders) | 1 | 0
Burning Sensation (Nervous system disorders) | 1 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 2 | 0
Cognitive Disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 16 | 1
Dizziness Postural (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 11 | 2
Headache (Nervous system disorders) | 24 | 3
Hypoaesthesia (Nervous system disorders) | 3 | 0
Lethargy (Nervous system disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 1 | 0
Mental Impairment (Nervous system disorders) | 1 | 0
Muscle Spasticity (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 14 | 2
Paraesthesia (Nervous system disorders) | 3 | 3
Peripheral Motor Neuropathy (Nervous system disorders) | 3 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 20 | 3
Peroneal Nerve Palsy (Nervous system disorders) | 0 | 1
Restless Legs Syndrome (Nervous system disorders) | 3 | 0
Seizure (Nervous system disorders) | 1 | 0
Sinus Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Taste Disorder (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 3 | 0
Vith Nerve Disorder (Nervous system disorders) | 0 | 1
Device Malfunction (Product Issues) | 1 | 0
Agitation (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 9 | 0
Confusional State (Psychiatric disorders) | 4 | 0
Depression (Psychiatric disorders) | 10 | 1
Emotional Disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 28 | 2
Irritability (Psychiatric disorders) | 3 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Personality Change (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 2 | 0
Bladder Discomfort (Renal and urinary disorders) | 1 | 0
Bladder Outlet Obstruction (Renal and urinary disorders) | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 6 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 4 | 2
Pollakiuria (Renal and urinary disorders) | 3 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 3 | 0
Urinary Hesitation (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 0
Urine Flow Decreased (Renal and urinary disorders) | 0 | 1
Urogenital Fistula (Renal and urinary disorders) | 1 | 0
Breast Calcifications (Reproductive system and breast disorders) | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 2 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 | 0
Genital Erythema (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Nipple Pain (Reproductive system and breast disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 2 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Symptom (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 1
Chronic Pigmented Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Nail Pigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 4 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 1
Rash Follicular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Mass (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0
Menopause (Social circumstances) | 1 | 0
Catheterisation Venous (Surgical and medical procedures) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 3 | 0
Flushing (Vascular disorders) | 12 | 1
Haematoma (Vascular disorders) | 1 | 0
Hot Flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 8 | 1
Hypotension (Vascular disorders) | 6 | 2
Pallor (Vascular disorders) | 1 | 0
Varicose Vein (Vascular disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT02951819/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT02951819/SAP_001.pdf